CLINICAL TRIAL: NCT03377322
Title: A Randomized Double-Blinded Placebo-Controlled Trial of Probiotics for Constipation in Parkinson's Disease
Brief Title: Trial of Probiotics for Constipation in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ProbioRCT
Record Dates: First submitted 2017-12-07; First posted 2017-12-19 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Placebo Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Probiotics capsules
  Interventions: Drug: Probiotic Capsule
- Placebo (Placebo Comparator): Placebo capsules containing maltodextrin
  Interventions: Drug: Placebo Capsule

INTERVENTIONS:
Drug: Probiotic Capsule — Probiotic - one capsule a day for four weeks
  Arms: Treatment
Drug: Placebo Capsule — Placebo - one capsule a day for four weeks
  Arms: Placebo

SUMMARY:
This is a double blinded randomised placebo controlled trial to evaluate the efficacy of probiotics in the treatment of constipation in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 to 80 years old
* Provision of written informed consent
* Diagnosis of PD made by a Neurologist using UK Brain Bank Criteria
* Fulfils criteria for functional constipation according to the Rome IV Criteria during in the preceding 6 months with frequency of bowel movements less than 3 times per week

Exclusion Criteria:

* Ingestion of probiotics in the preceding 4 weeks
* Use of antibiotics in the preceding 4 weeks
* History of gastrointestinal disorders or surgery
* Known or suspected allergy to probiotics
* Comorbidities that prevent reliable completion of study assessments
* Prior functional neurosurgery for PD or treatment with apomorphine infusion
* Recent initiation of dopaminergic medications in the preceding 3 months

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Change in frequency of bowel opening per week | Week 4 post randomisation
  Average number of bowel opening per week based on stool diary

SECONDARY OUTCOMES:
Change in stool consistency | Week 4 post randomisation
  Average stool consistency based on Bristol stool chart that was included in the stool diary
Change in constipation severity score | Week 4 post randomisation
  Total score of a constipation severity questionnaire adapted from ROME IV criteria for functional constipation. This scale evaluates the severity of five parameters related to constipation which include straining during defecation, lumpy or hard stools, sensation of incomplete evacuation, manual manoeuvres to facilitate defecations and spontaneous bowel movements per week. Each parameter is scored from 0 to 3, with 3 indicating the worst severity.
Change in patient's quality of life in relation to constipation | Week 4 post randomisation
  Total score of PAC-QOL questionnaire (Marquis et al, Scandinavian J of Gastroenterology 2008). This scale has a total of 28 items evaluating four different constructs related to quality of life which include worries/concerns, physical discomfort, psychosocial discomfort and patient's satisfaction. Each item is scored from 1 to 5, with 5 indicating the worst severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ai Huey Tan, MD,FRCP, Principal Investigator — University of Malaya
Locations (1):
- University of Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Todd CL, Johnson EE, Stewart F, Wallace SA, Bryant A, Woodward S, Norton C. Conservative, physical and surgical interventions for managing faecal incontinence and constipation in adults with central neurological diseases. Cochrane Database Syst Rev. 2024 Oct 29;10(10):CD002115. doi: 10.1002/14651858.CD002115.pub6. PMID 39470206
- [Derived] Tan AH, Lim SY, Chong KK, A Manap MAA, Hor JW, Lim JL, Low SC, Chong CW, Mahadeva S, Lang AE. Probiotics for Constipation in Parkinson Disease: A Randomized Placebo-Controlled Study. Neurology. 2021 Feb 2;96(5):e772-e782. doi: 10.1212/WNL.0000000000010998. Epub 2020 Oct 12. PMID 33046607